CLINICAL TRIAL: NCT01273935
Title: Dose-Dependent Effect of Early Antiplatelet Therapy in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Medical Faculty Ruhr-University Bochum, Dekanat der Medizinischen Fakultät, Forschungsreferat - FoRUM
Other Study IDs: MevesASS01
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Test the Efficacy of Antiplatelet Regimes in Acute Stroke
Keywords: Aspirin, Acute Cerebrovascular Ischemia, Platelet Function

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Responder: Responder versus Non-Responder as a result of platelet function test
- Non-Responder: According to the result of platelet function test

SUMMARY:
The aim of this study is to evaluate the low-response prevalence of early antiplatelet therapy and to test the influence of different aspirin dosages in patients with acute ischemic strokes (AIS).

DETAILED DESCRIPTION:
Antiplatelet agents are important therapeutic options in treating patients with acute ischemic strokes to prevent recurrent ischemic events or death. The aim of this study was to evaluate the low-response prevalence of early antiplatelet therapy and the influence of different aspirin dosages in patients with acute ischemic strokes (AIS).

ELIGIBILITY:
Inclusion Criteria:

* suspected acute cerebrovascular ischemic events and patients who were admitted to the stroke unit where antiplatelet therapy was initiated

Exclusion Criteria:

* severe liver disorders, current gastrointestinal disorders, congestive heart failure, life-threatening malignancies and a personal or family history of bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the stroke unit
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-01; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Result of platelet function test
  Aggregometry result of antiplatelet therapy

CONTACTS AND LOCATIONS:
Overall Officials: Saskia H Meves, MD, Principal Investigator — Department of Neurology, St. Josef - Hospital, Bochum, Germany
Locations (1):
- Department of Neurology, St. Josef - Hospital, Ruhr-University, Bochum, North Rhine-Westphalia, Germany